CLINICAL TRIAL: NCT03122236
Title: Combining tDCS and Neurorehabilitation to Treat Age-related Deficits of Mobility and Cognition: UPfront Walking Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB201602317 -N; R21AG053736 (NIH)
Record Dates: First submitted 2017-04-07; First posted 2017-04-20 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Mobility Limitation; Cognitive Impairment
MeSH Terms: conditions — Mobility Limitation; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will take part in a 6-week, 18-session neurorehabilitation led by qualified and trained study personnel. Participants will be randomized to one of three groups: 1) standard walking neurorehabilitation with sham tDCS ('standard/sham' group), 2) complex walking neurorehabilitation with sham tDCS ('complex/sham' group), or 3) complex walking neurorehabilitation with active anodal tDCS ('complex/active' group). Training logs will be maintained to gauge the content and intensity of training.
Who Masked: Participant, Investigator
Masking Description: To control for intensity, participants will maintain a rating of perceived exertion of 4 (moderate to strong) on the Borg Category/Ratio Scale during walking. Exertion will be adjusted by modifying walking speed and/or by modifying the rest time between walking bouts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard walking with Sham tDCS (Active Comparator): Neurorehabilitation of Standard Walking and Sham Transcranial Direct Current Stimulation (Sham tDCS)
  Interventions: Behavioral: Neurorehabilitation of Standard Walking; Device: Sham Transcranial Direct Current Stimulation (Sham tDCS)
- Complex walking with Sham tDCS (Active Comparator): Neurorehabilitation of Complex Walking and Sham Transcranial Direct Current Stimulation (Sham tDCS)
  Interventions: Behavioral: Neurorehabilitation of Complex Walking; Device: Sham Transcranial Direct Current Stimulation (Sham tDCS)
- Complex walking with Active tDCS (Active Comparator): Neurorehabilitation of Complex Walking and Active Transcranial Direct Current Stimulation (Active tDCS)
  Interventions: Behavioral: Neurorehabilitation of Complex Walking; Device: Active Transcranial Direct Current Stimulation (Active tDCS)

INTERVENTIONS:
Behavioral: Neurorehabilitation of Standard Walking — Neurorehabilitation is a behavioral therapeutic approach for enhancing the neural control of task performance by: Restoration of function, specificity of training, Sensory input to the nervous system, Intensity, Repetition and Progression of training. Neurorehabilitation of standard walking will focus on the use of typical steady state walking.
  Arms: Standard walking with Sham tDCS
Behavioral: Neurorehabilitation of Complex Walking — Neurorehabilitation is a behavioral therapeutic approach for enhancing the neural control of task performance by: Restoration of function, specificity of training, Sensory input to the nervous system, Intensity, Repetition and Progression of training. Neurorehabilitation of complex walking will focus on the use of walking tasks that require increased attention and executive functions. The following walking tasks will be used: over obstacles, navigating around obstacles, changing speeds, on soft surfaces (exercise mat), in dim lighting, while conversing with the therapist, up/down ramps and climbing/descending stairs.
  Arms: Complex walking with Active tDCS; Complex walking with Sham tDCS
Device: Sham Transcranial Direct Current Stimulation (Sham tDCS) — tDCS will be used to induce positive neuromodulation of frontal/executive circuits to make them more amenable to the "activity-dependent neuroplasticity" that is known to occur with behavioral neurorehabilitation. Specifically, tDCS may facilitate the efficacy of our walking neurorehabilitation intervention by strengthening the synaptic connections within the recruited circuits.
  Other Names: Soterix Direct Current Stimulator
  Arms: Complex walking with Sham tDCS; Standard walking with Sham tDCS
Device: Active Transcranial Direct Current Stimulation (Active tDCS) — tDCS will be used to induce positive neuromodulation of frontal/executive circuits to make them more amenable to the "activity-dependent neuroplasticity" that is known to occur with behavioral neurorehabilitation. Specifically, tDCS may facilitate the efficacy of our walking neurorehabilitation intervention by strengthening the synaptic connections within the recruited circuits.
  Other Names: Soterix Direct Current Stimulator
  Arms: Complex walking with Active tDCS

SUMMARY:
Loss of mobility and cognitive ability are serious conditions that threaten the independence of older adults. The objective of this study is to initiate a line of research to develop a novel therapeutic intervention to enhance both mobility and cognition via neuroplasticity of frontal/executive circuits.

DETAILED DESCRIPTION:
Frontal lobe dysfunction has been implicated as a factor contributing to gait deficits in some individuals with Alzheimer's disease, frontotemporal dementia and vascular dementia. There is a critical gap in knowledge about what therapeutic strategies are effective for maintaining or reinstating function in this critical brain region in order to preserve physical and cognitive health in older adults. The goal of our research is to develop a novel therapeutic intervention to enhance both mobility and cognition via neuroplasticity of frontal/executive control circuits. The Investigator will engage neuroplasticity of frontal circuits in two ways. The first is through neurorehabilitation with "complex walking tasks" (CWTs), such as obstacle crossing, obstacle avoidance and walking on non-uniform surfaces. CWTs are a potent behavioral approach for engaging prefrontal circuits. Furthermore, CWTs are crucial to successful ambulation in the home and community settings and therefore provide an ecologically valid therapeutic approach. The second approach that the Investigator will use to engage neuroplasticity of frontal circuits is anodal transcranial direct current stimulation (tDCS). Anodal tDCS is a safe, non-invasive neuromodulation technique. It has previously been shown to induce excitatory effects on brain tissue and, in single-session assessments, to improve performance during complex walking tasks. tDCS has also been shown to be an effective adjuvant for enhancing the effects of cognitive training. The objective of this study is to calculate effect size, establish variance of response and demonstrate feasibility of the experimental interventions in order to plan for a full scale clinical trial. Participants will include thirty older adults who demonstrate evidence of frontal/executive impairment. Participants will be randomized to one of three groups: 1) standard walking neurorehabilitation with sham tDCS ('standard/sham' group), 2) complex walking neurorehabilitation with sham tDCS ('complex/sham' group), or 3) complex walking neurorehabilitation with active anodal tDCS ('complex/active' group). Functional near infrared spectroscopy (fNIRS) will be used to explore intervention-induced changes in prefrontal cortical activity. Assessments will be conducted at baseline, post-treatment and 3-month follow up. The Investigator propose the following specific aims:

Specific Aim 1: Determine preliminary efficacy for recovery of mobility and cognitive function.

Specific Aim 2: Demonstrate feasibility/safety of tDCS as an adjuvant to rehabilitation.

Specific Aim 3: Explore the relationship between prefrontal activity and behavioral outcomes The data collected here will provide the information needed to justify and plan a future full scale clinical trial to assess the relative efficacy and underlying mechanisms of each intervention approach.

ELIGIBILITY:
Inclusion criteria

* preferred 10m walking speed < 1.0 m/s
* 40th-80th percentile rank (age and education corrected score) on NIH toolbox executive assessments: Card Sort Test and Flanker test
* willingness to be randomized to either intervention and to participate in all aspects of study assessment and intervention

Exclusion criteria

* contraindications to non-invasive brain stimulation and/or MRI including metal in the head, pacemaker, known abnormal cranial fissures/holes.
* difficulty communicating with study personnel
* uncontrolled hypertension at rest (systolic > 180 mmHg and/or diastolic > 100 mmHg)
* low vision that cannot be corrected by wearing glasses. Low visual will be operationally defined as visual acuity less than 20/70 on a standard eye chart, or difficulty performing complex walking tasks due to visual conditions affecting accurate navigation around and over obstacles (self-reported or observed by examiner).
* illiterate, due to the likelihood of difficulties performing some of the cognitive tasks
* non-English speaking, due to the likelihood of difficulties following instructions during therapy and during assessments
* use of medications that are know to modify tDCS effectiveness including those with anticholinergic, GABAergic, or glutamatergic properties, or sodium channel blockers
* clinical judgment of investigative team

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2021-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Clark, ScD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - HealthStreet, Gainesville, Florida
  - UF Institute on Aging, Gainesville, Florida
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chatterjee SA, Seidler RD, Skinner JW, Lysne PE, Sumonthee C, Wu SS, Cohen RA, Rose DK, Woods AJ, Clark DJ. Effects of Prefrontal Transcranial Direct Current Stimulation on Retention of Performance Gains on an Obstacle Negotiation Task in Older Adults. Neuromodulation. 2023 Jun;26(4):829-839. doi: 10.1016/j.neurom.2022.02.231. Epub 2022 Apr 8. PMID 35410769

RESULTS

PARTICIPANT FLOW:
Groups:
- Complex Walking With Active tDCS: Neurorehabilitation of Complex Walking and Active Transcranial Direct Current Stimulation (Active tDCS)
  Neurorehabilitation of Complex Walking: Neurorehabilitation is a behavioral therapeutic approach for enhancing the neural control of task performance by: Restoration of function, specificity of training, Sensory input to the nervous system, Intensity, Repetition and Progression of training. Neurorehabilitation of complex walking will focus on the use of walking tasks that require increased attention and executive functions. The following walking tasks will be used: over obstacles, navigating around obstacles, changing speeds, on soft surfaces (exercise mat), in dim lighting, while conversing with the therapist, up/down ramps and climbing/descending stairs.
  Acive Transcranial Direct Current Stimulation (Active tDCS): tDCS will be used to induce positive neuromodulation of frontal/executive circuits to make them more amenable to the "activity-dependent neuroplasticity" that is known to occur with behavioral neurorehabilitation. Specifically, tDCS may facilitate the efficacy of our walking neurorehabilitation intervention by strengthening the synaptic connections within the recruited circuits.
- Complex Walking With Sham tDCS: Neurorehabilitation of Complex Walking and Sham Transcranial Direct Current Stimulation (Sham tDCS)
  Neurorehabilitation of Complex Walking: Neurorehabilitation is a behavioral therapeutic approach for enhancing the neural control of task performance by: Restoration of function, specificity of training, Sensory input to the nervous system, Intensity, Repetition and Progression of training. Neurorehabilitation of complex walking will focus on the use of walking tasks that require increased attention and executive functions. The following walking tasks will be used: over obstacles, navigating around obstacles, changing speeds, on soft surfaces (exercise mat), in dim lighting, while conversing with the therapist, up/down ramps and climbing/descending stairs.
  Sham Transcranial Direct Current Stimulation (Sham tDCS): Sham tDCS is a placebo to Active tDCS.
- Standard Walking With Sham tDCS: Neurorehabilitation of Standard Walking and Sham Transcranial Direct Current Stimulation (Sham tDCS)
  Neurorehabilitation of Standard Walking: Neurorehabilitation is a behavioral therapeutic approach for enhancing the neural control of task performance by: Restoration of function, specificity of training, Sensory input to the nervous system, Intensity, Repetition and Progression of training. Neurorehabilitation of standard walking will focus on the use of typical steady state walking.
  Sham Transcranial Direct Current Stimulation (Sham tDCS): Sham tDCS is a placebo to Active tDCS.
Period: Overall Study
Arm/Group | Complex Walking With Active tDCS | Complex Walking With Sham tDCS | Standard Walking With Sham tDCS
Started | 7 | 6 | 7
Completed | 7 | 5 | 6
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Complex Walking With Active tDCS: Neurorehabilitation of Complex Walking and Transcranial Direct Current Stimulation (tDCS) dosage B
  Neurorehabilitation of Complex Walking: Neurorehabilitation is a behavioral therapeutic approach for enhancing the neural control of task performance by: Restoration of function, specificity of training, Sensory input to the nervous system, Intensity, Repetition and Progression of training. Neurorehabilitation of complex walking will focus on the use of walking tasks that require increased attention and executive functions. The following walking tasks will be used: over obstacles, navigating around obstacles, changing speeds, on soft surfaces (exercise mat), in dim lighting, while conversing with the therapist, up/down ramps and climbing/descending stairs.
  Active Transcranial Direct Current Stimulation (Active tDCS): tDCS will be used to induce positive neuromodulation of frontal/executive circuits to make them more amenable to the "activity-dependent neuroplasticity" that is known to occur with behavioral neurorehabilitation. Specifically, tDCS may facilitate the efficacy of our walking neurorehabilitation intervention by strengthening the synaptic connections within the recruited circuits.
- Complex Walking With tDCS Dosage A: Neurorehabilitation of Complex Walking and Sham Transcranial Direct Current Stimulation (Sham tDCS)
  Neurorehabilitation of Complex Walking: Neurorehabilitation is a behavioral therapeutic approach for enhancing the neural control of task performance by: Restoration of function, specificity of training, Sensory input to the nervous system, Intensity, Repetition and Progression of training. Neurorehabilitation of complex walking will focus on the use of walking tasks that require increased attention and executive functions. The following walking tasks will be used: over obstacles, navigating around obstacles, changing speeds, on soft surfaces (exercise mat), in dim lighting, while conversing with the therapist, up/down ramps and climbing/descending stairs.
  Sham Transcranial Direct Current Stimulation (tDCS): Sham tDCS is a placebo to Active tDCS
- Standard Walking With tDCS Dosage A: Neurorehabilitation of Standard Walking and Sham Transcranial Direct Current Stimulation (Sham tDCS)
  Neurorehabilitation of Standard Walking: Neurorehabilitation is a behavioral therapeutic approach for enhancing the neural control of task performance by: Restoration of function, specificity of training, Sensory input to the nervous system, Intensity, Repetition and Progression of training. Neurorehabilitation of standard walking will focus on the use of typical steady state walking.
  Sham Transcranial Direct Current Stimulation (tDCS): Sham tDCS is a placebo to Active tDCS
- Total: Total of all reporting groups
Arm/Group | Complex Walking With Active tDCS | Complex Walking With tDCS Dosage A | Standard Walking With tDCS Dosage A | Total
Number analyzed (Participants) | 7 | 6 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.4 (5.8) | 70.6 (5.2) | 73.7 (7.6) | 73.2 (6.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 15
  Male | 2 | 1 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 3 | 6
  White | 6 | 4 | 4 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Typical Walking Speed [Mean (Standard Deviation); unit: meters per second] | 0.94 (0.18) | 0.95 (0.15) | 0.97 (0.12) | 0.95 (0.16)

OUTCOME MEASURES:

1. Primary Outcome: Mobility: Figure-of-eight Walking Test (Figure-8 Walk Test)
Description: Time to complete a walking course at usual pace. The course is 15 feet in length and arranged as a Figure-8 pattern.
Time Frame: Change (value at 6 weeks minus value at baseline)
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Complex Walking With Active tDCS: Neurorehabilitation of Complex Walking and Transcranial Direct Current Stimulation (tDCS) dosage B
  Neurorehabilitation of Complex Walking: Neurorehabilitation is a behavioral therapeutic approach for enhancing the neural control of task performance by: Restoration of function, specificity of training, Sensory input to the nervous system, Intensity, Repetition and Progression of training. Neurorehabilitation of complex walking will focus on the use of walking tasks that require increased attention and executive functions. The following walking tasks will be used: over obstacles, navigating around obstacles, changing speeds, on soft surfaces (exercise mat), in dim lighting, while conversing with the therapist, up/down ramps and climbing/descending stairs.
  Transcranial Direct Current Stimulation (tDCS) dosage B: tDCS will be used to induce positive neuromodulation of frontal/executive circuits to make them more amenable to the "activity-dependent neuroplasticity" that is known to occur with behavioral neurorehabilitation. Specifically, tDCS may facilitate the efficacy of our walking neurorehabilitation intervention by strengthening the synaptic connections within the recruited circuits.
- Complex Walking With Sham tDCS: Neurorehabilitation of Complex Walking and Transcranial Direct Current Stimulation (tDCS) dosage A
  Neurorehabilitation of Complex Walking: Neurorehabilitation is a behavioral therapeutic approach for enhancing the neural control of task performance by: Restoration of function, specificity of training, Sensory input to the nervous system, Intensity, Repetition and Progression of training. Neurorehabilitation of complex walking will focus on the use of walking tasks that require increased attention and executive functions. The following walking tasks will be used: over obstacles, navigating around obstacles, changing speeds, on soft surfaces (exercise mat), in dim lighting, while conversing with the therapist, up/down ramps and climbing/descending stairs.
  Transcranial Direct Current Stimulation (tDCS) dosage A: tDCS will be used to induce positive neuromodulation of frontal/executive circuits to make them more amenable to the "activity-dependent neuroplasticity" that is known to occur with behavioral neurorehabilitation. Specifically, tDCS may facilitate the efficacy of our walking neurorehabilitation intervention by strengthening the synaptic connections within the recruited circuits.
- Standard Walking With Sham tDCS: Neurorehabilitation of Standard Walking and Transcranial Direct Current Stimulation (tDCS) dosage A
  Neurorehabilitation of Standard Walking: Neurorehabilitation is a behavioral therapeutic approach for enhancing the neural control of task performance by: Restoration of function, specificity of training, Sensory input to the nervous system, Intensity, Repetition and Progression of training. Neurorehabilitation of standard walking will focus on the use of typical steady state walking.
  Transcranial Direct Current Stimulation (tDCS) dosage A: tDCS will be used to induce positive neuromodulation of frontal/executive circuits to make them more amenable to the "activity-dependent neuroplasticity" that is known to occur with behavioral neurorehabilitation. Specifically, tDCS may facilitate the efficacy of our walking neurorehabilitation intervention by strengthening the synaptic connections within the recruited circuits.
Arm/Group | Complex Walking With Active tDCS | Complex Walking With Sham tDCS | Standard Walking With Sham tDCS
Number analyzed (Participants) | 7 | 5 | 6
seconds | 10.57 (1.93) | 9.58 (1.42) | 11.00 (2.00)

2. Secondary Outcome: Cognitive Composite Executive Score on EXAMINER Battery
Description: EXAMINER is an acronym for "Executive Abilities:Measures and Instruments for Neurobehavioral Evaluation and Research.
  EXAMINER is a battery of assessments that tests 7 domains of executive function separately and as a composite score. The composite score is based on Item Response Theory (logistic modeling) and ranges from a minimum value of -4 to a maximum value of 4. Higher scores indicate better performance.
Time Frame: Change (value at 6 weeks minus value at baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Complex Walking With Active tDCS | Complex Walking With Sham tDCS | Standard Walking With Sham tDCS
Number analyzed (Participants) | 7 | 5 | 6
units on a scale | -0.19 (0.74) | 0.29 (0.22) | 0.03 (0.96)

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Complex Walking With Sham tDCS: Neurorehabilitation of Complex Walking and Sham Transcranial Direct Current Stimulation (Sham tDCS)
  Neurorehabilitation of Complex Walking: Neurorehabilitation is a behavioral therapeutic approach for enhancing the neural control of task performance by: Restoration of function, specificity of training, Sensory input to the nervous system, Intensity, Repetition and Progression of training. Neurorehabilitation of complex walking will focus on the use of walking tasks that require increased attention and executive functions. The following walking tasks will be used: over obstacles, navigating around obstacles, changing speeds, on soft surfaces (exercise mat), in dim lighting, while conversing with the therapist, up/down ramps and climbing/descending stairs.
  Sham Transcranial Direct Current Stimulation (tDCS): Sham tDCS is a placebo to Active tDCS
- Standard Walking With Sham tDCS: Neurorehabilitation of Standard Walking and Sham Transcranial Direct Current Stimulation (Sham tDCS)
  Neurorehabilitation of Standard Walking: Neurorehabilitation is a behavioral therapeutic approach for enhancing the neural control of task performance by: Restoration of function, specificity of training, Sensory input to the nervous system, Intensity, Repetition and Progression of training. Neurorehabilitation of standard walking will focus on the use of typical steady state walking.
  Sham Transcranial Direct Current Stimulation (tDCS): Sham tDCS is a placebo to Active tDCS
Arm/Group | Complex Walking With Active tDCS | Complex Walking With Sham tDCS | Standard Walking With Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 1/7 | 2/6 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Complex Walking With Active tDCS (N=7) | Complex Walking With Sham tDCS (N=6) | Standard Walking With Sham tDCS (N=7)
kidney stones (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Complex Walking With Active tDCS (N=7) | Complex Walking With Sham tDCS (N=6) | Standard Walking With Sham tDCS (N=7)
Falling (no injury) (General disorders) | 1 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT03122236/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT03122236/ICF_001.pdf